CLINICAL TRIAL: NCT07237425
Title: A Safety, Efficacy and Pharmacokinetic Evaluation Study of Intralesional Ronkyla Plus Injection for the Treatment of Superficial Lipoma
Brief Title: Intralesional Ronkyla Plus Injection for the Treatment of Superficial Lipoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Glonova Pharma Co., Ltd (Industry)
Collaborators: T-TOP Clinical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDC003
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lipoma; Submental Fullness
Keywords: ATX-101; Ronkyla Plus
MeSH Terms: conditions — Lipoma | interventions — Saline Solution; Deoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Ronkyla Plus will be studied in four dose-escalating cohorts in Part I, with each subsequent cohort initiated only after a favorable safety profile has been observed in the first treatment cycle of the preceding cohort and the sponsor and the investigator determine that the trial can proceed. Part II will utilize a parallel study model where subjects with superficial lipoma(s) or submental fullness will be assigned to Ronkyla Plus or Kybella treatment cohort, respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Part I study will be conducted under double-blind conditions. All subjects, investigators and most of the study site staff will be blinded to the treatment assignment either at the time of randomization or later throughout the conduct of the study. In the meantime, the designated site staff responsible for IMP preparation and the designated CRO's data analysis team responsible for generating the randomization code list will be the only individuals unblinded to the treatment assignment.
  The Part II study will be conducted under open-label conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part I: Dose Level 1 (Experimental): 0.25 mL/cm2 of Ronkyla Plus (n=3), or placebo in equivalent injection volume/lipoma size (n=1) every 4 weeks for up to 6 treatments.
  Interventions: Drug: Ronkyla Plus; Drug: Placebo
- Part I: Dose Level 2 (Experimental): 0.5 mL/cm2 of Ronkyla Plus (n=3), or placebo in equivalent injection volume/lipoma size (n=1) every 4 weeks for up to 6 treatments.
  Interventions: Drug: Ronkyla Plus; Drug: Placebo
- Part I: Dose Level 3 (Experimental): 0.75 mL/cm2 of Ronkyla Plus (n=3), or placebo in equivalent injection volume/lipoma size (n=1) every 4 weeks for up to 6 treatments.
  Interventions: Drug: Ronkyla Plus; Drug: Placebo
- Part I: Dose Level 4 (Experimental): 1.0 mL/cm2 of Ronkyla Plus (n=3), or placebo in equivalent injection volume/lipoma size (n=1) every 4 weeks for up to 6 treatments.
  Interventions: Drug: Ronkyla Plus; Drug: Placebo
- Part II: Ronkyla Plus treatment (Experimental): Eligible subjects with a treatable superficial lipoma will receive a single treatment of Ronkyla Plus at the maximum tolerated dose determined in Part I and undergo a 16-day PK assessment.
  Interventions: Drug: Ronkyla Plus
- Part II: Kybella treatment (Active Comparator): Eligible subjects with submental fullness will receive a single treatment of Kybella at the maximum approved dose for a single session (100 mg) and undergo a 16-day PK assessment.
  Interventions: Drug: Kybella

INTERVENTIONS:
Drug: Ronkyla Plus — Ronkyla Plus is a new formulation of sodium deoxycholate lipolysis injection. It forms a hydrogel at the injection site.
  Arms: Part I: Dose Level 1; Part I: Dose Level 2; Part I: Dose Level 3; Part I: Dose Level 4; Part II: Ronkyla Plus treatment
Drug: Placebo — Normal saline for injection.
  Other Names: Normal saline
  Arms: Part I: Dose Level 1; Part I: Dose Level 2; Part I: Dose Level 3; Part I: Dose Level 4
Drug: Kybella — 10 mg/mL deoxycholic acid injection
  Other Names: deoxycholic acid; ATX-101
  Arms: Part II: Kybella treatment

SUMMARY:
This study aims to evaluate the safety, efficacy, and pharmacokinetics of Ronkyla Plus, a combinational drug that forms a hydrogel at the injection site, promising a better experience of lipolysis injection for the treatment of superficial lipoma. The study consists of a Part I dose-escalation study to investigate the drug's maximum tolerated dose (MTD) for this indication and a Part II study for evaluating its relative bioavailability in comparison to an FDA-approved lipolysis injection, Kybella.

DETAILED DESCRIPTION:
Part I is a randomized, double-blind, placebo-controlled, and sequential dose-escalation study. Eligible subjects will receive intralesional injections of Ronkyla Plus or placebo at a volume dependent on the size of their superficial lipoma, up to a maximum of 10 mL per treatment, at 28-day intervals for up to a maximum of 6 treatments. In the first treatment cycle, subjects will stay in hospital for 3 hours after treatment for evaluation of acute safety profile. Subjects will return to the hospital on Day 8 and Day 29 of each treatment cycle for safety profile evaluation.

Part II is an open-label, single-dose, 2-treatment, parallel study to evaluate the relative bioavailability of Ronkyla Plus injection in comparison with that of Kybella injection. Eligible, non-smoking males and females aged 18 to 65 with treatable superficial lipoma or submental fullness will be included in the study. Twenty (20) subjects for each target symptom, in a total of 40 subjects, are planned to be enrolled in the study to achieve at least 16 evaluable subjects in each treatment group. After screening, subjects will be assigned to Ronkyla Plus or Kybella treatment based on their symptoms and undergo a 16-day PK assessment.

For Ronkyla Plus injection, subject will receive a single intralesional treatment at the maximum tolerated dose (MTD) as determined in Part I. For Kybella injection, subject will receive the maximum dose approved for a single treatment (100 mg) in the submental area.

In the PK assessment period, subjects will visit the hospital in the mornings of Day 3 (48.0 h), Day 5 (96.0 h), Day 8 (168.0 h), Day 11 (240.0 h), and Day 15 (336.0 h), and two consecutive 24-hr PK blood samplings from Day -2 evening to Day 2 morning (pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0 h post-dose on Day 1~Day 2; same blood sampling time on Day -1~Day 1 without dosing). Two weeks after the end of the 16-day PK assessment period, subjects of Ronkyla Plus cohort will be eligible for up to 5 additional treatments of Ronkyla Plus for complete clearance of their target superficial lipomas, whereas subjects of Kybella cohort will be eligible for up to 5 additional treatments of Ronkyla (10.56 mg/mL SDC injection approved in Taiwan for submental fullness treatment, pharmaceutical equivalent of Kybella) for improvement of their submental fullness.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adults aged 18 to 65 years, inclusive.
2. One or more superficial lipomas, based on clinical diagnosis, which are accessible for treatment and assessment, are quantifiable along at least 2 perpendicular diameters, and have the following characteristics:

   * History of slow growth followed by dormancy, and stable for at least 6 months.
   * Greatest length by greatest perpendicular width between 1 and 10 square centimeters, inclusive.
   * Discrete, oval to rounded in shape, not hard or attached to underlying tissue.
   * Located on the trunk, arms, legs, or neck
   * Needle biopsy core tissue sample histological analysis results consistent with a diagnosis of lipoma.

   OR, sufficient submental fat for injection of 100 mg Kybella in the judgment of the investigator (Part II Kybella cohort only)
3. Body mass index (BMI): BMI between 22 to 30 (normal, overweight and slight obese).
4. History of stable body weight, in the judgment of the investigator, for at least 6 months before enrollment.
5. The health status is assessed by the investigator as "normal healthy" based on required screening assessments.
6. Females of childbearing potential must have a negative human chorionic gonadotropin (hCG) test result within 28 days before enrollment and agree to use a highly effective method of contraception from enrollment up to the study end, such as:

   * Intrauterine device
   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with the inhibition of ovulation (oral, intravaginal, or transdermal)
   * Progestogen-only hormonal contraception associated with the inhibition of ovulation (oral, injectable, intrauterine, or implantable)
   * Tubal ligation
   * Vasectomized male partner
   * Sexual abstinence

   Female subject being postmenopausal for at least 1 year or surgically sterile is considered to be of no childbearing potential.
7. Able and willing to comply with scheduled clinic visits and clinical trial procedures.
8. Capable of understanding and giving signed informed consent form after full discussion of the research nature of the treatment and its risk and benefits with the investigator/ designee of the sponsor.

Exclusion Criteria:

1. History of surgical treatment for the target superficial lipoma or submental area (Part II Kybella cohort only).
2. Current infection or wound near the target superficial lipoma or the submental area (Part II Kybella cohort only).
3. History of diabetes.
4. Allergic to excipients of Ronkyla Plus or Kybella (Part II Kybella cohort only)
5. A result on coagulation tests (prothrombin time, activated partial thromboplastin time) obtained within 28 days before enrollment that indicates the presence of any clinically significant bleeding disorder (subjects being treated with antiplatelet therapy or anticoagulants could be enrolled after 7-day washout period):

   * Prothrombin time > 20 seconds.
   * Activated partial thromboplastin time > 60 seconds.
   * INR > 3.
6. Any ongoing medical condition with significant risk of bleeding
7. Evidence of any serious active infections, COVID 19, severe uncontrolled cardiac, renal, hepatic, pulmonary or other systemic disease, significant medical or psychiatric condition, known seropositivity to HIV/HBV/HCV, or clinically significant laboratory findings that would, in the investigator's judgment, make the subject inappropriate for the study.
8. Administration of an investigational drug within 30 days prior to enrollment.
9. Administration of a COVID-19 vaccine within 30 days prior to enrollment.
10. Abnormal hepatic and renal functions; hematologic changes at screening:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 X upper limit of normal (ULN).
    * Total bilirubin > 1.5 X ULN.
    * Serum creatinine > 1.5 X ULN.
    * Hemoglobin < lower limit of normal (LLN).
    * Platelets ≤ 100.000/mm³.
11. Current malignancy of any organ system or a history within 5 years.
12. Subjects who, in the opinion of the investigator, are not likely to complete the trial for whatever reason.

Part I & Part II Ronkyla Plus cohort specific exclusion criteria:

1. History of any medical condition contraindicated or not recommended for aspirin use including active peptic ulcer disease, asthma, gout, uncontrolled hypertension.
2. Taking any medication contraindicated or not recommended for concomitant use with aspirin within 7 days prior to enrollment.
3. Allergic to Aspirin, salicylates, or non-steroidal anti-inflammatory drugs (NSAIDs).
4. The target lipoma warrants surgical removal per the investigator's judgement (e.g., for confirming its pathology).

Part I dose level 2 and 4 cohorts & Part II specific exclusion criteria:

1. History of alcohol or drug abuse within the past year prior to Day 1.
2. History of smoking or use of nicotine-containing product within 6 months prior to Day 1.
3. Donation or significant loss of blood (480 mL or more) within 60 days prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Part I: Incidence of all adverse events | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure
Part I: Incidence of all serious adverse events | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure
Part I: Incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥2 bone marrow toxicities | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. CTCAE version 5.0 (Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening, Grade 5: Death)
Part I: Incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥2 cardiac toxicities | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. CTCAE version 5.0 (Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening, Grade 5: Death)
Part I: Change from baseline in vital signs | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Measurement of blood pressure (including systolic blood pressure and diastolic blood pressure, unit: mmHg; pulse rate, unit: beats/mins; respiratory rate, unit: times/min; body temperature, unit: degree Celsius)
Part I: Change from baseline in physical and weight measurement | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Physical examination includes: general appearance and weight (kg), HEENT (head, eyes, ears, nose, and throat), mouth, skin, neck (including thyroid), lymph nodes, spine, cardiovascular system, gastrointestinal system, nervous system, musculoskeletal system, mental status.
Part I: Change from baseline in Comprehensive Metabolic Panel blood test | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Blood test for: albumin, blood urea nitrogen, calcium, carbon dioxide, chloride, creatinine, glucose, potassium, sodium, total bilirubin and protein, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase
Part I: Change from baseline in Complete blood count test | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Blood test includes: hemoglobin, hematocrit, red blood cell, white blood cell (neutrophils, band %, segment %, eosinophils, basophils, lymphocytes, and monocytes), platelet count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin
Part I: Change from baseline in lipid profile. | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Blood test includes: total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglyceride.
Part I: Change from baseline in thyroid test. | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Blood test includes: triidothyronine, thyroxine, and thyroid-stimulating hormone.
Part I: Change from baseline in urinalysis | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Measurement includes: pH, protein, occult blood, leukocyte, glucose, ketones, bilirubin, urobilinogen, nitrite, clinical microscopy.
Part I: Change from baseline in inflammation evaluation. | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Test includes: c-reactive protein, erythrocyte sedimentation rate
Part I: Change from baseline in coagulation function. | 7 months (Part I); 1 month (Part II)
  Also a Part II Secondary Outcome Measure. Blood test includes: prothrombin time, activated partial thromboplastin time
Part II: Baseline-adjusted area under the plasma concentration-time curve over a 24-hour period (AUC0-24) of deoxycholic acid | 16 days
  PK values on Day -1~Day 1 (pre-dosing) will be subtracted from PK values on Day 1 ~Day 15 (post-dosing)
Part II: Baseline-adjusted area under the curve from zero to time infinity (AUC0-inf) of deoxycholic acid | 16 days
  PK values on Day -1~Day 1 (pre-dosing) will be subtracted from PK values on Day 1 ~Day 15 (post-dosing)
Part II: Baseline-adjusted peak plasma concentration (Cmax) of deoxycholic acid | 16 days
  PK values on Day -1~Day 1 (pre-dosing) will be subtracted from PK values on Day 1 ~Day 15 (post-dosing)
Part II: Baseline-adjusted time to maximum concentration (Tmax) of deoxycholic acid | 16 days
  PK values on Day -1~Day 1 (pre-dosing) will be subtracted from PK values on Day 1 ~Day 15 (post-dosing)
Part II: Baseline-adjusted elimination half-life (T1/2) of deoxycholic acid | 16 days
  PK values on Day -1~Day 1 (pre-dosing) will be subtracted from PK values on Day 1 ~Day 15 (post-dosing)
Part II: Baseline-adjusted, dose-normalized area under the plasma concentration-time curve over a 24-hour period (AUC0-24) | 16 days
  Baseline-adjusted PK values will be divided by the injected dose of deoxycholic acid
Part II: Baseline-adjusted, dose-normalized area under the curve from zero to time infinity (AUC0-inf) of deoxycholic acid | 16 days
  Baseline-adjusted PK values will be divided by the injected dose of deoxycholic acid
Part II: Baseline-adjusted, dose-normalized peak plasma concentration (Cmax) of deoxycholic acid | 16 days
  Baseline-adjusted PK values will be divided by injected dose of deoxycholic acid
Part II: Baseline-adjusted, dose-normalized time to maximum concentration (Tmax) of deoxycholic acid | 16 days
  Baseline-adjusted PK values will be divided by the injected dose of deoxycholic acid.
Part II: Baseline-adjusted, dose-normalized elimination half-life (T1/2) of deoxycholic acid | 16 days
  Baseline-adjusted PK values will be divided by the injected dose of deoxycholic acid

SECONDARY OUTCOMES:
Percentage of subjects with "complete" or "almost complete" clearance of the target superficial lipoma at the end of Cycle 2 (Part I only) | 2 months
  At screening, 1 target superficial lipoma will be selected for treatment. Lipoma will be measured in ≥ 2 dimensions (longest length, perpendicular width, and height if possible) using both digital calipers and ultrasound imaging.
  Almost complete clearance is defined as ≥ 90% reduction in surface area of the target superficial lipoma
Percentage of subjects with "complete" or "almost complete" clearance of the target superficial lipoma at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort
Percentage of subjects with "complete" clearance of the target superficial lipoma at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort
Percentage of subjects with "almost complete" clearance of the target superficial lipoma at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort
Percentage reduction in size of the target superficial lipoma at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort
Percentage of subjects having their target superficial lipoma rated by the investigator as 0 or 1 point on the investigator's lipoma morphology assessment scale at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort.
  At screening, the beginning/end of each treatment cycle, and the end of study, the investigator will use a 4-point scale of 0-3 to rate the morphology of subjects' target lipomas where 0= Not palpable, 1=Not visible, barely palpable, 2=Visible upon palpation, and 3=Clearly visible, easily palpable. A score of 0 to 1 indicates favorable morphological changes of the target lipoma following treatment(s).
Percentage of subjects having their target superficial lipoma rated by the investigator with ≥2 points improvement on the investigator's lipoma morphology assessment scale at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort. Investigator's lipoma morphology assessment scale where 0 = not palpable; 1 = not visible, barely palpable; 2 = visible upon palpation; 3 = clearly visible, easily palpable. The percentage of subjects having their target superficial lipomas assessed by the investigator on the scale as follows: 0 or 1 point; with ≥ 2 points improvement from baseline; with ≥ 1 point improvement from baseline.
Percentage of subjects having their target superficial lipoma rated by the investigator with ≥1 point improvement on the investigator's lipoma morphology assessment scale at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort. Investigator's lipoma morphology assessment scale where 0 = not palpable; 1 = not visible, barely palpable; 2 = visible upon palpation; 3 = clearly visible, easily palpable. The percentage of subjects having their target superficial lipomas assessed by the investigator on the scale as follows: 0 or 1 point; with ≥ 2 points improvement from baseline; with ≥ 1 point improvement from baseline.
Percentage of subjects being satisfied with treatment outcome at the end of each treatment cycle and end of study | 7 months (Part I); 1 month (Part II)
  Days 29, 57, 85, 113, 141, 169, 197 for Part I; Day 29 for Part II Ronkyla Plus cohort.
  Satisfaction assessment will be performed independently by subjects using a 5-point scale where 0 = worsen, 1 = no response, 2 = moderate response, 3 = good response, and 4 = excellent response. A score of 3 or 4 qualifies for a satisfactory treatment outcome.
Injection site pain rated by subjects on a 0-10 numeric rating scale (NRS) at 1 hour and 1 week after each treatment | 25 weeks (Part I); 1 week (Part II)
  Days 1, 8, 29, 36, 57, 64, 85, 92, 113, 120, 141, 148 for Part I; Days 1, 8 for Part II Ronkyla Plus cohort.
  At approximately 1 hour after each treatment, and at the 1-week follow-up visit for each treatment, subjects will be asked to rate their injection site pain using a 0-10 numeric rating scale (NRS) where 0 = no pain and 10 = most severe pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiu Yen, MD, Principal Investigator — Cathay General Hospital
Locations (2):
- Taiwan (2):
  - Cathay General Hospital, Taipei, Da'an District
  - Cathay General Hospital Sijhih Branch, New Taipei City, Sijhih District

IPD SHARING:
Plan to Share IPD: No